CLINICAL TRIAL: NCT03126032
Title: Early Detection of Glycocalyx Damage in Emergency Room Patients
Acronym: EDGE
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 001
Record Dates: First submitted 2017-02-20; First posted 2017-04-24 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Sepsis; SIRS
Keywords: Sepsis; SIRS; Glycocalyx; Glycocheck™-System; Infection
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with suspected sepsis: Patients presenting in the Emergency Room (ER) with the clinical suspicion of infection/sepsis.
  Evaluation of the glycocalyx damage with the use of GlycoCheck™-System, as well as blood sample at presentation, day 1 and day 7 of their hospital stay.
  Interventions: Other: GlycoCheck™-System
- Non-Sepsis Patients: Patients presenting in the Emergency Room with other conditions apart from infection/sepsis.
  Evaluation of their sublingual glycocalyx and blood sample for further microbiologic and laboratory analysis at presentation.
  Interventions: Other: GlycoCheck™-System
- Healthy Individuals: Evaluation of their sublingual glycocalyx and blood sample for further microbiologic and laboratory analysis at presentation.
  Interventions: Other: GlycoCheck™-System

INTERVENTIONS:
Other: GlycoCheck™-System — Consecutive, sublingual measurements of endothelial glycocalyx with GlycoCheck™-System will be obtained at presentation, as well as during the inpatient treatment of the patients with suspected sepsis.
  Blood sample will be drawn in all groups at time of assessment. Besides that, in patients with suspected sepsis blood samples will be drawn for further microbiologic and laboratory analysis at day 1 and day 7 of their hospital stay.

SUMMARY:
Aim of the study is to evaluate to what extent a glycocalyx damage measured in the ER in patients presenting with sepsis correlates with their clinical course and if it can be used as a clinical stratification tool and mortality predictor.

The study will focus on the changes of the microcirculation and how they correlate with the macrocirculation, as well as microbiologic parameters. In the study will participate ca. 300 patients with sepsis, as well as 30 patients without sepsis and 30 healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected sepsis

* Adult patients presenting to the ER with the clinical suspicion of infection
* Indication for hospital admission

Patients without sepsis

* Adult patients presenting to the ER with other conditions apart from sepsis/infection.

Healthy individuals

* Adult healthy individuals.

Exclusion Criteria (for all groups):

* Underage persons
* Pregnant women
* Oral mucosal injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non consecutive patients presenting in the ER of the University Hospital in Muenster, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of glycocalyx thickness with clinical course. | At time of presentation in the ER.
  Glycocalyx thickness measured with the use of GlycoCheck System (Perfused Boundary Region - PBR, in µm) will be correlated with patients' clinical course (e.g. with the use of SOFA score - pts.).

SECONDARY OUTCOMES:
Correlation of glycocalyx thickness with major events. | Hospital stay, an expected average of 4 weeks.
  Glycocalyx thickness (PBR, in µm) will be correlated with patients΄ major events (dialysis, intubation, ICU admission, death)
Correlation of glycocalyx thickness with 90-day mortality. | Up to 90 days.
  Glycocalyx thickness (PBR, in µm) will be correlated with patients΄ 90-day mortality.
Correlation of glycocalyx thickness with subsequent organ failure. | Hospital stay, an expected average of 4 weeks.
  Glycocalyx thickness (PBR, in µm) will be correlated with subsequent organ failure (e.g. kidney, lung, circulation).

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kümpers, MD, Principal Investigator — University Muenster
Locations (1):
- Universitiy Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description of GlycoCheck™- System — http://microvascular.com/wp-content/uploads/2015/01/MicroVascular-Health-Solutions-Glycocalyx-White-Paper.pdf